CLINICAL TRIAL: NCT00932412
Title: A Randomized Phase II Study of Clofarabine / Intermediate-Dose Cytarabine (CLARA)Versus High-Dose Cytarabine (HDAC) as Consolidation in Younger Patients With Newly-Diagnosed Acute Myeloid Leukemia (AML).
Brief Title: The CLARA Study From the Acute Leukemia French Association (ALFA 0702 Trial)
Acronym: CLARA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006.456/50
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Younger Patients with Newly-Diagnosed Acute Myeloid Leukemia (AML).
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLARA (Experimental): Clofarabine / Intermediate-Dose Cytarabine (CLARA) with G-CSF given during each sequence of chemotherapy in order to increase the blast priming.
  Interventions: Drug: CLARA
- HDAC (Active Comparator): High-Dose Cytarabine (HDAC) with G-CSF given during each sequence of chemotherapy in order to increase the blast priming.
  Interventions: Drug: HDAc

INTERVENTIONS:
Drug: CLARA — Clofarabine 30 mg/m2/day IV (2h) on days 2 to 6 (administered as a 2h infusion in 250 ml of 0.9% normal saline solution) Cytarabine 1 g/m2/day intravenous (2h) 4 hours later on days 1 to 5 (administered as a 2h infusion in 250 ml of 5% dextrose in water) G-CSF 5 microg/kg/day intravenous from day 1 to day 6 (administered as a 30 mn infusion in 20 ml of dextrose 5% in water)
  Arms: CLARA
Drug: HDAc — Cytarabine 3 g/m2/12h intravenous (3h) on days 1, 3, 5 (administered as a 3h infusion in 250 ml of 5% dextrose in water) G-CSF 5 microg/kg/day intravenous from day 1 to day 5 (administered as a 30 mn infusion in 20 ml of dextrose 5% in water)
  Arms: HDAC

SUMMARY:
This study is a phase II randomized multicenter study. Patients will be enrolled at time of diagnosis and will receive one or two cycles of induction chemotherapy. Patients, without indication of intensification by allogeneic stem cell transplantation and/or without HLA (Human Leukocyte Antigen)-compatible donor, who attain a CR after one or two cycles of induction chemotherapy, will be eligible for the study Clofarabine / Intermediate-Dose Cytarabine (CLARA)versus High-Dose Cytarabine (HDAC)and will be randomized between 3 courses of CLARA chemotherapy and 3 courses of HDAC chemotherapy as consolidation.

We will compare efficacy and toxicity among the two arms.

DETAILED DESCRIPTION:
Because of the results of our former trial (ALFA-9802) [Thomas, 2005], chemotherapy will be combined in each arm with G-CSF (Granulocyte Colony-Stimulating Factor) given during each sequence of chemotherapy in order to increase the blast priming.

ELIGIBILITY:
Inclusion Criteria at registration:

1. Age 18 years or more and less than 60 years
2. With:

   A morphologically proven diagnosis of AML according to the WHO classification, cytogenetically (standard karyotype, FISH-MLL) and molecularly (FLT3, CEBPA, NMP1) defined.
3. ECOG (Eastern Cooperative Oncology Group) performance status 0 to 2.
4. Have adequate renal and hepatic function as indicated by the following laboratory values:

   * Creatinine clearance (calculated by the cockcroft and Gault method) ≥ 40mL/min;
   * AST (Aspartate amino transférase) and ALT (Alanine Amino Transférase ) < or = 2.5N; total bilirubin < or = 2N (unless related to the underlying disease).
5. Cardiac function determined by radionuclide or echography within normal limits.
6. Women of child-bearing potential (i.e. women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods, and must have a negative serum or urine pregnancy test within 2 weeks prior the beginning treatment on this trial.
7. Must be able and willing to give written informed consent.
8. The subject must be covered by a social security system.

Exclusion Criteria at registration:

1. Patients with AML with favorable risk cytogenetics: M3-AML; CBF-AML including t(8:21), inv(16), or t(16;16) AML.
2. Ph-positive AML.
3. AML following diagnosed myeloproliferation or patient with prior history of MDS known for more than 3 months
4. Prior treatment with chemotherapy or radiotherapy for another tumor.
5. Prior tumor, if not stable for at least two years, except in-situ carcinoma and skin carcinoma
6. Compromised organ function judged to be lifethreatening by the Investigator.
7. Positive serology for HIV (Human Immunodeficiency Virus), HBV (Hepatitis B Virus) and HBC (Hepatitis C Virus)(except post vaccination)
8. Uncontrolled active infection of any kind or bleeding. Patients with infections who are under active treatment with antibiotics and whose infections are controlled may be entered to the study.
9. Other active malignancy.
10. Patients concurrently receiving any other standard or investigational treatment for their leukemia, with the exception of hydroxyurea.

INCLUSION CRITERIA AT RANDOMIZATION

1. Patients with either in first CR/CRp after the first induction course or in first CR/CRp after salvage therapy.
2. ECOG performance status 0 to 2.
3. AST and ALT < or = 2.5N; total bilirubin < or = 2N.
4. Creatinine clearance ≥40mL/min (calculated by the cockcroft and Gault method or by MDRD (see http://nephron.org/cgi-bin/MDRD_GFR/cgi)
5. Patient without HLA identical donor.

   EXCLUSION CRITERIA AT RANDOMIZATION
6. Patients belonging to the intermediate 1 risk group (CEBPA+ or NPM1+ without Flt3-ITD) in CR/CRp after the first induction course. These patients will go out of the study and receive consolidation cycles based on HD-AraC (Aracytine).
7. Known central nervous system involvement with AML.
8. Uncontrolled active infection of any kind or bleeding.
9. Compromized organ function judged to be lifethreatening by the Investigator.
10. Patient with HLA identical donor identified.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 735 (Actual)
Dates: Start 2009-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
DFS (disease free survival) following first remission achievement (CR : Complete Remission or CRp : Complete Remission but platelet count < 100 x109/L) in younger patients with intermediate-risk or unfavorable-risk AML. | 2 years
  As all these patients are eligible for allogenic stem cell transplantation in first remission if they have a donor and the comparison of interest primarily concerns non-transplanted patients, it is planned: 1) to exclude patients with an identified donor; 2) to adjust Relapse Free survival (RFS) comparison on the interaction with stem cell transplantation in first remission; and 3) to censure at transplant time the patients allografted before disease progression after randomization (late donor identification) as sensitivity analysis.

SECONDARY OUTCOMES:
• Safety profile of CLARA versus HDAC consolidation courses | 2 years
  All toxicity encountered during therapy will be evaluated according to the CTC expanded Common Toxicity Criteria and causal relationship to investigational products will be reported.
  Serious Adverse Events encountered 3 MONTHS after the last cycle of study chemotherapy (induction/salvage/CLARA/HDAC), whether or not ascribed to the study, will be recorded in the Serious Adverse Event form.
• Possible predictors to response | 2 years
  Possible predictors to response: with respect to cytogenetics risk groups and mutational status: FLT3 (Fms-like tyrosine kinase 3), MLL (myeloid/ lymphoid or mixed-lineage leukemia), CEBPA (CCAAT / enhancer binding protein α) and NPM(Nucleophosmin))
• MRD (Minimal Residual Disease) level | 2 years
  Evaluation of MRD in patients with AML in clinical remission is a potentially useful tool for assessing the risk of relapse and guiding further therapeutic decisions. Once an aberrant pattern is identified at diagnosis, it will serve as a "patient-specific probe" to be used, with standard triple/quadruple labelling, to track residual disease longitudinally. Bone marrow and peripheral blood samples for MRD evaluation will be collected at fixed time points:
  * End of induction in patients achieving CR/CRp.
  * End of consolidation 3.
  * Every 6 months during follow-up for 2 years.
• Overall cumulative incidence of relapse | 120 days
• Overall survival (OS) | 2 years
  OS will be defined as the time from diagnosis to death or last contact with the patient

CONTACTS AND LOCATIONS:
Overall Officials: Xavier THOMAS, MD, Principal Investigator — Hospices Civils de Lyon
Locations (34):
- France (34):
  - Hôpital Sud - CHU Amiens, Amiens
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - Hôpital Victor Dupouy, Argenteuil
  - Hôpital Avicenne - bobigny, Bobigny
  - Centre Hospitalier Boulogne/Mer, Boulogne / Mer
  - Hôpital Clemenceau - chu Caen, Caen
  - Centre Hospitalier René Dubos, Cergy-Pontoise
  - HIA Percy, Clamart
  - Hôpital de Corbeil, Corbeil
  - Hôpital Mondor, Créteil
  - Hôpital Dubocage, Dijon
  - Centre Hospitalier Dunkerque, Dunkirk
  - Hôpital Michallon, Grenoble
  - Centre Hospitalier Versailles, Le Chesnay
  - Centre Hospitalier Schaffner, Lens
  - Hôpital Huriez, Lille
  - CHU Dupuytren, Limoges
  - Institut Paoli-Calmette, Marseille
  - Centre Hospitalier Meaux, Meaux
  - CHU - Hôtel Dieu, Nantes
  - Centre A. Lacassagne, Nice
  - Hôpital Archet 1, Nice
  - Hôpital St Louis, Paris
  - Pitié-Salpetrière, Paris
  - Paris Necker, Paris
  - Hôpital Haut Lévêque, Pessac
  - Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital V. Provo, Roubaix
  - Centre Henri Becquerel - CHRU ROUEN, Rouen
  - Centre Hospitalier Huguenin, Saint-Cloud
  - Hôpital Purpan, Toulouse
  - Centre Hospitalier Valenciennes, Valenciennes
  - CHU de Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Michallet M, Sobh M, Morisset S, Deloire A, Raffoux E, de Botton S, Caillot D, Chantepie S, Girault S, Berthon C, Bertoli S, Lepretre S, Leguay T, Castaigne S, Marolleau JP, Pautas C, Malfuson JV, Veyn N, Braun T, Gastaud L, Suarez F, Schmidt A, Gressin R, Bonmati C, Celli-Lebras K, El-Hamri M, Ribaud P, Dombret H, Thomas X, Bergeron A. Antifungal Prophylaxis in AML Patients Receiving Intensive Induction Chemotherapy: A Prospective Observational Study From the Acute Leukaemia French Association (ALFA) Group. Clin Lymphoma Myeloma Leuk. 2022 May;22(5):311-318. doi: 10.1016/j.clml.2021.10.011. Epub 2021 Oct 25. PMID 34895843
- [Background] Fenwarth L, Thomas X, de Botton S, Duployez N, Bourhis JH, Lesieur A, Fortin G, Meslin PA, Yakoub-Agha I, Sujobert P, Dumas PY, Recher C, Lebon D, Berthon C, Michallet M, Pigneux A, Nguyen S, Chantepie S, Vey N, Raffoux E, Celli-Lebras K, Gardin C, Lambert J, Malfuson JV, Caillot D, Maury S, Ducourneau B, Turlure P, Lemasle E, Pautas C, Chevret S, Terre C, Boissel N, Socie G, Dombret H, Preudhomme C, Itzykson R. A personalized approach to guide allogeneic stem cell transplantation in younger adults with acute myeloid leukemia. Blood. 2021 Jan 28;137(4):524-532. doi: 10.1182/blood.2020005524. PMID 32871585
- [Background] Hirsch P, Lambert J, Bucci M, Deswarte C, Boudry A, Lambert J, Fenwarth L, Micol JB, Terre C, Celli-Lebras K, Thomas X, Dombret H, Duployez N, Preudhomme C, Itzykson R, Delhommeau F. Multi-target measurable residual disease assessed by error-corrected sequencing in patients with acute myeloid leukemia: An ALFA study. Blood Cancer J. 2024 Jun 13;14(1):97. doi: 10.1038/s41408-024-01078-8. PMID 38871702